CLINICAL TRIAL: NCT04119700
Title: Fistulectomy With Primary Sphincter Reconstruction vs. Muco-muscular Endorectal Advancement Flap in the Treatment of High Transsphincteric Anal Fistulas
Brief Title: Fistulectomy and Primary Sphincter rEconstruction vs. endorectaL Advancement Flap in the Treatment of High Anal Fistulas
Acronym: SELF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 070819
Record Dates: First submitted 2019-10-06; First posted 2019-10-08 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Anal Fistula
Keywords: fistulectomy; fistula; advancement flap; transsphincteric fistula; sphincteroplasty; primary sphincter reconstruction; high fistula; endorectal flap
MeSH Terms: conditions — Rectal Fistula; Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Muco-muscular endorectal advancement flap (Active Comparator): After fistulectomy a muco-muscular endorectal advancement flap is mobilised and fixed to anoderma
  Interventions: Procedure: Muco-muscular endorectal advancement flap after fistulectomy
- Primary sphincter reconstruction (Experimental): After fistulectomy the defect in anal sphincters is closed
  Interventions: Procedure: Primary sphincter reconstruction after fistulectomy

INTERVENTIONS:
Procedure: Muco-muscular endorectal advancement flap after fistulectomy — After fistulectomy muco-muscular flap of the rectal wall will be mobilized. The muscular defect is sutured with separate interrupted sutures (Vicryl / Polysorb 2/0, 0/0, 3/0). The muco-muscular flap is fixed to the anoderm without tension by interrupted sutures (Vicryl / Polysorb 4/0). The wound of the perianal area is not sutured.
  Arms: Muco-muscular endorectal advancement flap
Procedure: Primary sphincter reconstruction after fistulectomy — Fistulectomy will be performed. The affected gland is visualized and removed. If there are secondary extensions, they are excised also. Sphincter defect with stitches (suture material Vicryl / Polysorb 2/0, 0/0, 3/0) with restoration of the anal canal profile (suturing of the anodermal-skin border). The skin is not suturing.
  Arms: Primary sphincter reconstruction

SUMMARY:
The optimal method of surgical treatment of complex anorectal fistulas has not been found yet.

The aim of this study is to compare two techniques in treatment of high anorectal fistulas. This study purpose to demonstrate that the fistulectomy with dissection from 1/3 to 2/3 of the height of the sphincter complex with primary suturing is technically simpler, equally effective and safe in comparison with muco-muscular endorectal advancement flap.

DETAILED DESCRIPTION:
Anorectal fistula is a common proctological disease with prevalence between 8.6 and 10 per 100,000 population. Surgical treatment of complex anorectal fistulas has two main objectives: preventing the recurrence of the disease and preserving the anal continence. The optimal principle of management of patients with anorectal fistulas includes a comprehensive preoperative examination with the definition of the architectonics of the fistulous tract, the identification of the internal fistulous opening, the elimination of additional tracts and cavities.

Many methods are used for high anorectal fistula's treatment, but the optimal strategy has not been found yet.

Nowadays, the conventional sphincter-preserving operation for the treatment of complex anorectal fistulas is advancement rectal flap. In addition, plastic with a full-thickness flap in comparison with a mucosal flap was associated with less reccurence rate (10% and 40% respectively), and was accompanied by manifestation of incontinence symptoms, increased with the thickness of the flap.

About 20 years ago, in an attempt to reduce high level of incontinence, the primary reconstruction of sphincters after fistulotomy was proposed; however, this technique is still debated.

According to reports, dissection of more than 1/3 of the sphincter increases the incidence of postoperative incontinence. However, fistulectomy with primary suturing of the sphincter defect allows to improve the function of anal continence and is recommended for patients with initial incontinence after previous surgical interventions.

The studie's aim is comparison between two techniques in treatment of high anorectal fistulas. This study purpose to demonstrate that the fistulectomy with dissection from 1/3 to 2/3 of the height of the sphincter complex with primary suturing is technically simpler, equally effective and safe in comparison with muco-muscular endorectal advancement flap.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's consent to participate in the study
2. Patient's consent for surgery
3. High transsphincteric anorectal fistula, involving from 1/3 to 2/3 of the height of the sphincter according to the both MRI and intraoperative revision
4. Cryptoglandular fistulas
5. The absence of incontinence before the operation in accordance with the classification CCFF-IS
6. Preoperative MR-diagnostics before the operation

Exclusion Criteria:

1. Refuse of the patient to participate in the study.
2. Low transsphincteric (involving less than 1/3 of the height of the sphincter according to MRI), intersphincteric, extrasphincteric fistula of the rectum.
3. Recurrent fistula.
4. Rectovaginal or rectourethral fistula.
5. Anal incontinence (Appendix 2).
6. Pregnancy.
7. Inflammatory bowel disease (confirmed endoscopically and morphologically).
8. Patients with immunodepression (i.e. HIV)
9. The presence of an acute purulent process in the perianal area.
10. Anterior anorectal fistula in female.
11. The inability to perform MRI of the pelvic organs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2017-11-04 (Actual); Primary Completion 2020-02-20 (Estimated); Study Completion 2020-03-07 (Estimated)

PRIMARY OUTCOMES:
Incontinence rate | 1 day - 1 year
  The frequency of incontinence after the operation in accordance with the classification CCFF-IS (Cleveland Clinic Florida Faecal Incontinence Score). 0 points - total continence, 24 points - complete incontinence.

SECONDARY OUTCOMES:
Pain intencity | 1 day, 7 day, 14 day, 30 day
  The severity of pain in the postoperative period according to VAS score (visual analogue pain scale). Interpretation of values: no pain (0 points), mild pain (1-4 points), moderate pain (5-9 points), severe pain (10 points).
Recurrence rate | 1 day - 1 year
  The frequency of recurrence of the disease in the comparison groups during the observation period.
Wound healing | 30 day - 90 day
  The duration of wound healing in the perianal area and anus
Overall quality of life | assessed after surgery: 14 day, 1 month, 3 month, 6 month, 1 year
  Assessed with patient-reported questionnaire SF-36 (Short-form 36 Questionnaire). A total score in each of 8 sections will be calculated and transformed into a 0-100 scale with a score of zero equivalent to maximum disability and a score of 100 equivalent to no disabilityusing the SF-36 questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Tsarkov, Prof, Principal Investigator — Russian Society of Colorectal Surgeons
Locations (1):
- Clinic of Colorectal and Minimally Invasive Surgery, Moscow, Russia